CLINICAL TRIAL: NCT01567865
Title: A Clinical Trial in Healthy Infants to Assess Lot-to-lot Consistency of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine and Non-inferiority With Respect to an Earlier Product.
Brief Title: Lot-to-lot Consistency Trial of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JEV05 (VAC004)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Reference Lot (Active Comparator): Lot of Vaccine produced in existing facility
  Interventions: Biological: Vaccine produced in existing facility
- New Lot #1 (Experimental): First lot of vaccine produced in new facility
  Interventions: Biological: Vaccine produced in new facility
- New Lot #2 (Experimental): Second lot of vaccine produced in new facility
  Interventions: Biological: Vaccine produced in new facility
- New Lot #3 (Experimental): Third lot of vaccine produced in new facility
  Interventions: Biological: Vaccine produced in new facility

INTERVENTIONS:
Biological: Vaccine produced in existing facility — Live attenuated Japanese encephalitis vaccine SA 14-14-2 (LJEVac) produced in the existing facility by the Chengdu Institute of Biological Products (CDIBP), Chengdu, China
  Arms: Reference Lot
Biological: Vaccine produced in new facility — Live attenuated Japanese encephalitis vaccine SA 14-14-2 (LJEVac) produced in the new facility by the Chengdu Institute of Biological Products (CDIBP), Chengdu, China
  Arms: New Lot #1; New Lot #2; New Lot #3

SUMMARY:
The proposed study is a four-arm double-blind randomized controlled single center trial to evaluate, by examining post-vaccination seroprotection titers, the lot-to-lot consistency of three lots of Japanese Encephalitis live attenuated SA 14-14-2 vaccine (LJEVac) manufactured in a new good manufacture practice (GMP) facility, and to establish non-inferiority of the new vaccine in comparison to a single lot of the same vaccine manufactured in the existing facility. The study aimed to enroll a total of 1,000 Bangladeshi infants aged 10 to 12 months. In addition to providing immunogenicity data, this study provided local safety data of JE live attenuated SA 14-14-2 vaccine among Bangladeshi children. This is the first step to secure licensure for this life-saving vaccine in Bangladesh as well as provide data to support WHO prequalification of JE live attenuated SA 14-14-2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Infant's parent(s) or legal guardian(s) willing to provide signed informed consent.
* Healthy infants aged 10 to 12 months at enrolment residing in Matlab Health and Demographic Surveillance System (HDSS) intervention area who have completed all doses of Expanded Programme on Immunization (EPI) immunizations at least 4 weeks prior to enrolment: Bacillus Calmette-Guerin vaccine (BCG), Diphtheria-pertussis-tetanus vaccine (DPT), Hepatitis B (HBV), Haemophilus influenzae type (Hib), oral polio vaccine (OPV) and measles

Exclusion Criteria:

* Acute medical illness with or without fever within the last 72 hours or an axillary temperature (≥ 37.5°C ) at the time of vaccination.
* Use of antibiotics or antipyretics within the last 72 hours prior to enrolment.
* Severely or moderately malnourished infants (<-3 Z score).
* History of prematurity (< 36 weeks of pregnancy).
* Underlying medical condition such as failure to thrive, inborn errors of metabolism, bronchopulmonary dysplasia, or any major congenital abnormalities requiring surgery or chronic treatment.
* History of serious chronic disease (e.g., cardiac, renal, neurologic, metabolic, rheumatologic, hematologic, or bleeding disorder).
* Known or suspected impairment of immunologic function.
* History of documented or suspected encephalitis or meningitis.
* History of seizures, including history of febrile seizures, or any other neurologic disorder.
* History of JE infection.
* Prior receipt of a JE vaccine.
* Received measles vaccine within 4 weeks prior to, or scheduled to receive a vaccination during, the conduct of this trial.
* Prior or anticipated receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy within 6 weeks of administration of the study vaccine.
* Serious adverse reactions (e.g. urticaria, angioedema, shock, breathlessness following vaccination or any life threatening condition) with any previous EPI vaccine.
* Unable to attend the scheduled visits or comply with the study procedures.
* Enrolled in another clinical trial involving any therapy.
* Any condition that in the opinion of the investigator, would pose a health risk to the child, or interfere with the evaluation of the study objectives.

Ages: 10 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 818 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, MD, Principal Investigator — ICCDR,B
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

RESULTS

PARTICIPANT FLOW:
Period: Enrolled and Vaccinated (Day 0)
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
Started | 163 | 220 | 211 | 224
Completed | 163 | 220 | 211 | 224
Not Completed | 0 | 0 | 0 | 0
Period: Evaluated for Immunogenicity
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
Started | 163 | 220 | 211 | 224
Completed | 146 | 195 | 192 | 194
Not Completed | 17 | 25 | 19 | 30
Not completed — Sero+ for anti-JEV at Visit 1 | 0 | 1 | 3 | 2
Not completed — Missing blood sample | 17 | 24 | 16 | 28

BASELINE CHARACTERISTICS:
Population: Per-protocol population
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3 | Total
Number analyzed (Participants) | 146 | 195 | 192 | 194 | 727
Age, Continuous [Mean (Standard Deviation); unit: months] | 10.8 (.68) | 10.9 (.73) | 10.8 (.65) | 10.9 (.7) | 10.9 (.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 100 | 92 | 98 | 366
  Male | 70 | 95 | 100 | 96 | 361
Region of Enrollment [Number; unit: participants]
  Bangladesh | 146 | 195 | 192 | 194 | 727

OUTCOME MEASURES:

1. Primary Outcome: Number/Percentage of Subjects With Demonstrated Seroprotection
Description: Seroprotection was defined as a serum antibody titer equal to or greater than 1:10, as measured by Plaque reduction neutralization test (PRNT). The end point for neutralization was the highest dilution of serum reducing the number of plaques by 50%, compared with a negative serum control.
  In 2004, a group of experts under the leadership of the WHO recommended that seroprotection (SP) against JEV be defined as a neutralizing anti-JEV antibody serum titer ≥1:10 as determined by PRNT [Hombach et al. 2005]. Accordingly, a titer of ≥1:10 was adopted as an indicator of seroprotection in this study.
Time Frame: 28 days post-vaccination
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Groups:
- All New Lots: All subjects receiving vaccine from the new facility (Lot 1, 2, or 3)
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3 | All New Lots
Number analyzed (Participants) | 146 | 195 | 192 | 194 | 581
Participants
  Seroprotection | 126 | 160 | 154 | 164 | 478
  No seroprotection | 20 | 35 | 38 | 30 | 103
Statistical Analysis 1: Comparison: New Lot #1 vs New Lot #2; Null hypotheses: each new lot does not differ in seroprotection (SP) rates among each other by more than 10%. Slower than anticipated enrollment resulted in a smaller number of subjects with antibody response data for analysis. Consequently, additional power estimates were made in anticipation of the occurrence of smaller sample sizes. With a total study population of only 772 subjects, the power of the study to test lot-to-lot consistency declined from 90% to 85%; Test type: Equivalence — The 3 lots of new GMP facility LJEVac would be considered equivalent (i.e., the SP does not differ between lots by ≥10%) if all 3 null hypotheses are rejected, and the alternate hypotheses are accepted; Mean Difference (Net) = 1.84, 95% CI 2-sided [-5.97 to 9.66]
Statistical Analysis 2: Comparison: New Lot #1 vs New Lot #3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided; The 95% CI for the difference in rates is calculated based on the Newcombe-Wilson method without continuity correction; Mean Difference (Net) = -2.48, 95% CI 2-sided [-9.92 to 4.98]
Statistical Analysis 3: Comparison: New Lot #2 vs New Lot #3; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -4.33, 95% CI 2-sided [-11.94 to 3.31]
Statistical Analysis 4: Comparison: Reference Lot vs All New Lots; Null hypothesis: reference lot vs. Lot 1, 2, and 3 combined do differ in seroprotection (SP) rates among each other by more than 10%. Slower than anticipated enrollment resulted in a smaller number of subjects with antibody response data for analysis. Consequently, additional power estimates were made in anticipation of the occurrence of smaller sample sizes. The power of the study to test non-inferiority of the combined new lots compared to the reference lot dropped from 99% to 87%; Test type: Non-Inferiority — The new GMP facility lots will be considered non-inferior (i.e., equivalent) to the existing facility lot if the null hypothesis is rejected and the alternate hypothesis is accepted; p < 0.05, t-test, 2 sided; The 95% CI for the difference in rates is calculated based on the Newcombe-Wilson method without continuity correction; Mean Difference (Net) = -4.03, 95% CI 2-sided [-9.74 to 3.1]

2. Primary Outcome: Geometric Mean Titers (GMT)
Description: Geometric Mean Titers of Neutralizing anti-JEV antibody
Time Frame: 28 days post-vaccination
Population: Per-Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3 | All New Lots
Number analyzed (Participants) | 146 | 195 | 192 | 194 | 581
titer | 77.3 [59.6 to 100.4] | 52.8 [42.9 to 65.1] | 53.4 [42.4 to 67.2] | 62.8 [50.3 to 78.4] | 56.2 [49.5 to 63.8]

3. Secondary Outcome: Number/Percentage of Subjects With an Immediate Solicited Local or Systemic Reactogenicity Event (RE)
Description: Subjects were monitored for the following adverse events and categorized as events almost certainly related to receipt of the vaccine:
  Redness Swelling Tenderness Dyspnea Cyanosis Loose Stools Vomiting Convulsion Fever (37 degrees Celsius or greater, axillary) Hives (urticaria) Angioedema
Time Frame: Within 30 minutes of vaccination
Population: All study subjects receiving vaccine were included in this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
Number analyzed (Participants) | 163 | 220 | 211 | 224
Participants
  Any immediate RE | 0 | 6 | 5 | 2
  No immediate RE | 163 | 214 | 206 | 222

4. Secondary Outcome: Number/Percentage of Subjects With a Solicited Local or Systemic Reactogenicity Event Within 7 Days After Vaccination
Description: Collected by a home visit to observe the subject and interview his/her parent or guardian occurrence and severity of solicited injection site reactogenicity events (REs) related to vaccination and solicited systemic REs or other AEs that might or might not be related to the prior receipt of vaccine
Time Frame: Within 7 days of vaccination
Population: All subjects receiving the vaccine were assessed for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
Number analyzed (Participants) | 163 | 220 | 211 | 224
Participants
  Any RE | 51 | 75 | 81 | 61
  No RE | 112 | 145 | 130 | 163

5. Secondary Outcome: Number/Percentage of Subjects With Other Adverse Events (AE) During the Study
Description: Adverse events other than solicited reactogenicities were obtained through review of medical history when subject returned to clinic. They were graded for severity and rated by the PI for possible relationship to vaccination throughout the 28 days study period.
Time Frame: Between 7 and 28 days of vaccination
Population: All subjects receiving the vaccine were evaluated for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
Number analyzed (Participants) | 163 | 220 | 211 | 224
Participants
  Any AE | 60 | 84 | 92 | 77
  No AE | 103 | 136 | 119 | 147

ADVERSE EVENTS:
Time Frame: 28 days post-vaccination
Description: Adverse events other than solicited reactogenicities within the time frame. If the parent/guardian failed to come on day 28, a maximum of 4 days was allowed for follow-up.
Arm/Group | Reference Lot | New Lot #1 | New Lot #2 | New Lot #3
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/220 | 0/211 | 0/224
Serious Adverse Events (participants affected / at risk) | 2/163 | 4/220 | 4/211 | 0/224
Other Adverse Events (participants affected / at risk) | 60/163 | 84/220 | 92/211 | 77/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Lot (N=163) | New Lot #1 (N=220) | New Lot #2 (N=211) | New Lot #3 (N=224)
Severe pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Dysentery (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute watery diarrhea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Acute gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Lot (N=163) | New Lot #1 (N=220) | New Lot #2 (N=211) | New Lot #3 (N=224)
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 13 | 15 | 21 | 8
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 15 | 17 | 9
Injection site erythema (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0
Injection site pain (Gastrointestinal disorders) | 5 | 4 | 3 | 5
Injection site swelling (General disorders) | 1 | 1 | 2 | 0
Irritability (General disorders) | 7 | 9 | 8 | 6
Pain (General disorders) | 1 | 1 | 4 | 5
Pyrexia (General disorders) | 40 | 56 | 61 | 53
Swelling (General disorders) | 0 | 0 | 2 | 1
Tenderness (General disorders) | 7 | 5 | 6 | 10
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 8 | 3 | 4
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 36 | 27 | 31 | 31
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Crying (Nervous system disorders) | 13 | 11 | 12 | 11
Somnolence (Nervous system disorders) | 1 | 4 | 1 | 2
Insomnia (Psychiatric disorders) | 9 | 6 | 11 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 18 | 19 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 3 | 4
Rhinorhhea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 5 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritis generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Lower than anticipated rates of enrollment across all groups made it necessary to analyze antibody response data in smaller samples than initially planned. This adversely influenced the precision of all estimates (i.e., resulted in broader 95% CIs)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No